CLINICAL TRIAL: NCT05007535
Title: Tissue Characterization and Primary Percutaneous Coronary Intervention Guidance Using Intravascular Ultrasound
Acronym: SPECTRUM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Acist Medical Systems (Industry); MicroPort CRM (Industry)
Responsible Party: Principal Investigator, Joost Daemen, Principal Investigator, Erasmus Medical Center
Other Study IDs: SPECTRUM
Record Dates: First submitted 2021-04-21; First posted 2021-08-16 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: ST Elevation Myocardial Infarction; Acute Myocardial Infarction; Coronary Artery Disease; Percutaneous Coronary Intervention; Intravascular Ultrasound; Thrombus
Keywords: Invasive Coronary Imaging
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Coronary Artery Disease; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- HD-IVUS-guided primary PCI: Prospective, single arm, observational

SUMMARY:
This prospective, single arm, observational cohort study is designed to assess the safety and efficacy of (high-definition) intravascular ultrasound (HD-IVUS) as guidance for primary percutaneous coronary intervention (PCI) and to assess culprit lesion plaque characteristics and thrombus morphology in patients with ST-elevation myocardial infarction (STEMI).

Objectives:

* To assess clinical outcomes after IVUS-guided primary PCI in STEMI patients.
* To assess IVUS-guided optimization in STEMI patients.
* To assess culprit lesion plaque characteristics in STEMI patients with HD-IVUS.
* To assess and quantify thrombus in STEMI patients with HD-IVUS.
* To explore HD-IVUS derived predictors for clinically relevant aspiration thrombectomy.

DETAILED DESCRIPTION:
The SPECTRUM study is an investigator-initiated, single-center, prospective, single arm, observational cohort study investigating the safety and efficacy of (HD)-IVUS as guidance for primary PCI in 200 patients with STEMI. This study enables the assessment of culprit lesion plaque characteristics and thrombus morphology with a 40-60 MHz HD-IVUS catheter.

All study patients will have a protocolized pre-intervention IVUS pullback directly after recanalization (so before any lesion preparation, i.e. balloon dilatation, aspiration thrombectomy or stent placement) and a post-intervention IVUS pullback. Subsequently, if IVUS-guided optimization is performed, a final pullback is highly recommended and considered as the post-optimization IVUS pullback.

The primary study outcomes are target vessel failure at 12 months and incidence of IVUS-guided optimization. More information on outcome measures is provided in the section below.

ELIGIBILITY:
Inclusion Criteria:

* Native coronary artery culprit lesion, angiographically
* Culprit vessel reference diameter ≥ 2.25 mm, angiographically

Exclusion Criteria:

* Cardiogenic shock
* Presentation > 12 hours after symptom onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with ST-elevation myocardial infarction eligible for primary percutaneous coronary intervention.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-02-02 (Estimated); Study Completion 2023-02-02 (Estimated)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) | 12 Months
  A composite of cardiac death, target vessel myocardial infarction and clinically driven target vessel revascularization
IVUS-guided optimization | Procedural
  Incidence of IVUS-guided additional balloon dilatation or stent placement after angiographically successful PCI

SECONDARY OUTCOMES:
TVF | 30 Days
  A composite of cardiac death, target vessel myocardial infarction and clinically driven target vessel revascularization
Major Adverse Cardiovascular Events (MACE) | 30 Days
  A composite of all-cause mortality, any myocardial infarction and repeat revascularization
Major Adverse Cardiovascular Events (MACE) | 12 Months
  A composite of all-cause mortality, any myocardial infarction and repeat revascularization
Individual Components of TVF and MACE | 30 Days
  Individual components of the composite endpoints
Individual Components of TVF and MACE | 12 months
  Individual components of the composite endpoints
Major Intraprocedural Complications | Procedural
  Including type C-F dissections, perforations, slow flow or no-reflow, major side branch occlusion (> 2 mm)
Angiographic Endpoints | Procedural
  Including final TIMI flow and final myocardial blush grade
IVUS endpoints (continuous) | Procedural
  At least the following continuous variables will be assessed for the first 100 patients with sufficient HD-IVUS pullbacks:
  * Minimal lumen area
  * Thrombus containing frames
  * Thrombus maximum angle
  * Minimal stent area
  Structured analysis of the HD-IVUS pullbacks will be performed with dedicated invasive imaging analysis software.
IVUS endpoints (categorical) | Procedural
  At least the following categorical variables will be assessed for the first 100 patients with sufficient HD-IVUS pullbacks:
  * Plaque rupture
  * Convex calcium (nodule)
  * Thrombus type
  * Plaque type
  * Thrombus protrusion
  * Underexpansion
  * Edge dissection
  * Hematoma
  * High plaque burden at stent edges
  * Residual focal lesion
  * Malapposition
  Structured analysis of the HD-IVUS pullbacks will be performed with dedicated invasive imaging analysis software.

CONTACTS AND LOCATIONS:
Overall Officials: Joost Daemen, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groenland FTW, Ziedses des Plantes AC, Neleman T, Scoccia A, Ligthart JMR, Witberg KT, Mahmoud KD, Nuis RJ, den Dekker WK, Wilschut JM, Diletti R, Zijlstra F, Van Mieghem NM, Daemen J. Culprit lesion plaque characterization and thrombus grading by high-definition intravascular ultrasound in patients with ST-segment elevation myocardial infarction. Catheter Cardiovasc Interv. 2023 Aug;102(2):191-199. doi: 10.1002/ccd.30699. Epub 2023 May 26. PMID 37232425
- [Derived] Groenland FTW, Mahmoud KD, Neleman T, Ziedses des Plantes AC, Scoccia A, Ligthart J, Witberg KT, Nuis RJ, den Dekker WK, Wilschut JM, Diletti R, Zijlstra F, Kardys I, Cummins P, Van Mieghem NM, Daemen J. Tissue characterisation and primary percutaneous coronary intervention guidance using intravascular ultrasound: rationale and design of the SPECTRUM study. Open Heart. 2022 Apr;9(1):e001955. doi: 10.1136/openhrt-2021-001955. PMID 35437257